CLINICAL TRIAL: NCT06013046
Title: Wheelchair User Physical Activity Training Intervention to Enhance Cardiometabolic Health (WATCH): A Community-based Randomized Control Trial
Brief Title: Wheelchair User Physical Activity Training Intervention to Enhance Cardiometabolic Health
Acronym: WATCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kerri Morgan, Assistant Professor of Occupational Therapy and Neurology, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202209017; R01HD111022 (NIH)
Record Dates: First submitted 2023-06-02; First posted 2023-08-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Physical Disability
Keywords: Occupational Therapy; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensity-controlled physical activity training (IPAT) (Active Comparator): A group provided education on physical activity recommendations for people with disabilities, access to a community-based accessible gym, and an intensity-controlled 14-week one-on-one supervised physical activity training intervention.
  Interventions: Behavioral: Intensity-controlled physical activity training (IPAT)
- Education and Access (EA) (Placebo Comparator): A group provided education on physical activity recommendations for people with disabilities and access to a community-based accessible gym in order to independently complete a 14-week physical activity program.
  Interventions: Behavioral: Education and Access (EA)

INTERVENTIONS:
Behavioral: Intensity-controlled physical activity training (IPAT) — The IPAT group will receive 40 (90 minute) one-on-one, intensity-controlled, exercise sessions by trained staff over 14 weeks. The initial 2-week period will include dedicated education on topics including physical activity guidelines and the benefits of achieving them, the feeling of moderate-to-vigorous physical activity intensity levels, and the appropriate exercises for achieving desired intensity levels. Tailored sessions will be created for each participant based on their physical fitness, goals, preferred exercise equipment and results from their baseline assessment. Each session can include vitals, pain assessment, warm-up, aerobic training, strength exercises and a cool-down. The participants will be monitored to ensure they are achieving at least 150 minutes of moderate-to-vigorous intensity physical activity weekly. Heart rate and actigraphy monitors will be worn during sessions to capture exercise intensity data. The overall goal is to improve cardiorespiratory fitness.
  Arms: Intensity-controlled physical activity training (IPAT)
Behavioral: Education and Access (EA) — The EA group will receive an initial 60 minute educational session, during which they will receive information on the adapted exercise equipment in the Orthwein Center, education on the physical activity guidelines and the health benefits of achieving them, and access to the Orthwein Center accessible gym. They will then complete a 14-week independent workout program with the goal of meeting physical activities guidelines. They will have access to Orthwein Center staff to help with minimal setup and guidance, but sessions will be self-directed. Heart rate and actigraphy monitors will be worn during sessions to capture exercise intensity data. Participants will be asked to complete a log for each session to report pain, details of the activities they completed during their workout, the RPE for each activity, and how long each activity lasted.
  Arms: Education and Access (EA)

SUMMARY:
The goal of the study is to improve cardiometabolic health outcomes for wheelchair users and identify strategies for achieving sufficient physical activity intensity during bouts of structured physical activity.

DETAILED DESCRIPTION:
Wheelchair users have a higher risk for obesity and cardiometabolic health-related diseases compared to persons without a disability and remain one of the most sedentary populations in the United States. Engaging wheelchair users in physical activity levels following the current recommendations to achieve cardiometabolic health-related changes requires tailoring and supports in an accessible community environment, but it is unclear if a community-based physical activity intervention that also prioritizes intensity levels is best to improve cardiometabolic health. This project will determine the effects and implementation outcomes of a community-based, intensity-controlled aerobic and strength training intervention on the cardiometabolic health of wheelchair users and will significantly advance public health knowledge of how to engage wheelchair uses in physical activity to reverse or prevent cardiometabolic health-related disease.

The aims of the study are to:

1. Compare the effectiveness of the intensity-controlled physical activity training (IPAT) group to the education and access (EA) group for improving cardiometabolic-related health outcomes.
2. Identify barriers and facilitators to wheelchair users engaging in physical activity at a community-based accessible gym.
3. Examine the moderators (i.e., age, race, gender, duration of disability, wheelchair type, and physical function) and mediators (ie., self-efficacy, motivation, and barriers/facilitators) of the proposed intervention to understand for whom and how the intervention was effective.

A hybrid I RCT will be conducted. One hundred and ten individuals with a physical disability requiring the use of a wheelchair will be recruited. Each participant will be randomized into either a 14-week IPAT group (n=54) or a 14-week EA group (n=54). Participants' cardiorespiratory, body composition, metabolic blood chemistries and strength will be assessed baseline (T1) and post intervention (T2).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Has a physical disability requiring the use of a wheelchair (includes manual wheelchairs, motorized wheelchairs, motor-assisted wheelchairs, and electric scooters)
* Ability to attend weekly exercise sessions in person
* Ability to independently move one or both upper extremities
* Has participated in no more than 60 minutes of moderate-intensity physical activity per week in the past month
* English-speaking
* Able to provide informed consent
* Ability to complete a valid V02max score with 2 attempts

Exclusion Criteria:

* Determination by their physician to be medically unstable
* Has had cardiovascular complications within the past year or unstable heart disease
* Currently receiving medical treatment for an acute injury
* Presence of a stage IV pressure injury
* Currently pregnant or suspect pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
VO2max - Cardiorespiratory Fitness change (Max Oxygen Consumption Change in ml/kg/min) | Baseline and up to 3 weeks post intervention
  VO2max will be measured in ml/kg/min using a portable, breath-by-breath metabolic system with an optoelectronic reader, as well as reliable highly linear and rapid response O2 and CO2 sensors (COSMED K5, COSMED: The Metabolic Company, Chicago, IL). This testing will be completed while the participant performs a graded-exercise test on a crank ergometer (SCIFIT PRO2, Life Fitness, Tulsa, OK). The protocol involves a 3-minute warm-up followed by a standard ramp-up protocol which is typically completed in 8-12 minutes, and a subsequent 5-minute recovery phase.

SECONDARY OUTCOMES:
DEXA - Body Composition Overall Body Fat Change (kg) | Baseline and up to 3 weeks post intervention
  Participants will undergo body composition assessment via DEXA (General Electric Lunar iDXA), which is commonly used in research due to its precision and safety.
DEXA - Body Composition Overall Lean Mass Change (kg) | Baseline and up to 3 weeks post intervention
  Participants will undergo body composition assessment via DEXA (General Electric Lunar iDXA), which is commonly used in research due to its precision and safety.
Metabolic blood chemistries (fasting glucose and insulin) - Insulin Resistance Change (mg/dL) | Baseline and up to 3 weeks post intervention
  Participants will fast 8-10 hours prior to blood draw. Blood draws will be completed to determine both fasting glucose and fasting insulin. These results will then be used to figure the HOMA-IR score, which is an insulin resistance score in mg/dL .
Brachial artery reactivity test (BART) - Endothelial function change (%) | Baseline and up to 3 weeks post intervention
  Participants will undergo a BART via ultrasound. The test will measure flow-mediated dilation and endothelium independent dilation of the brachial artery using a high-resolution transducer on the Vivid E95, E9, Vivid IQ (portable) or Vivid I (portable) systems. Brachial artery flow-mediated vasodilation correlates with measures of coronary artery endothelial function and can predict future adverse coronary events.

OTHER OUTCOMES:
PROMIS - Change in Pain Intensity (Short Form 3a) | Baseline and up to 3 weeks post intervention
  The Pain Intensity instruments assess how much a person hurts. The pain intensity short forms are not disease specific and assess pain intensity over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "Had no pain (1)" to "very severe (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.
PROMIS - Change in Fatigue (Short Form 8a) | Baseline and up to 3 weeks post intervention
  The Fatigue item banks assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely impacts one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue and the impact of fatigue. The fatigue short forms are not disease specific and assess fatigue over the past seven days. PROMIS instruments are scored using item-level calibrations. Each question is answered using a 5-point Likert scale from "not at all (1)" to "very much (5)". Calculate a summed score and then use the applicable PROMIS score conversion table to translate the total raw score into a T-score.
  The seven domains are scored individually, and the single pain intensity item is reported as its raw score.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri A Morgan, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States